CLINICAL TRIAL: NCT00182390
Title: A Randomized Controlled Trial of Two Hemoglobin Thresholds for Transfusion in Newborns <1000g Birth Weight
Brief Title: Premature Infants in Need of Transfusion (PINT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTMG-2001-PINT; CIHR MCT-41549; CIHR MCT-58455
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Anemia of Prematurity
Keywords: ELBW premature infants; neonatal transfusion; bronchopulmonary dysplasia; periventricular leukomalacia; ventriculomegaly; retinopathy of prematurity
MeSH Terms: conditions — Anemia; Bronchopulmonary Dysplasia; Leukomalacia, Periventricular; Hydrocephalus; Retinopathy of Prematurity | interventions — Erythrocyte Transfusion

INTERVENTIONS:
Procedure: Red blood cell transfusion

SUMMARY:
Hypothesis: That a high hemoglobin threshold for transfusion in extremely low birth weight (ELBW) infants is associated with a lower rate of survival without severe morbidity (defined as one or more of retinopathy of prematurity, bronchopulmonary dysplasia, or periventricular leukomalacia/ventriculomegaly).

Primary Objective: To determine whether either a liberal or more restrictive threshold of hemoglobin level for red cell transfusion in ELBW infants is safer, by randomizing to either a high transfusion hemoglobin threshold or a low transfusion hemoglobin threshold.

Follow-up at a corrected age of 18 months represents a conventional age at which to first assess neurodevelopmental outcomes, and to predict long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* birth weight <1000g
* postnatal age <48 hours
* no transfusion beyond first 6 hours of life
* estimated gestational age of 30 completed weeks or less

Exclusion Criteria:

* infant considered non-viable by attending physician
* infant has cyanotic congenital heart disease
* infant's parents known to be opposed to blood transfusion
* either parent has hemoglobinopathies or congenital anemias
* infant has hemolytic disease
* infant has severe acute hemorrhage, severe shock, severe sepsis with coagulopathy or requires peri-operative transfusion
* prior treatment with or intention to treat with erythropoietin

Max Age: 48 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 424
Dates: Start 2001-02; Primary Completion 2003-02 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Combined mortality or survival to tertiary hospital discharge without severe morbidity (BPD, severe ROP or brain injury) | neonatal phase
Combined mortality or survival with neurodevelopmental disability (non-ambulatory cerebral palsy, blindness, deafness, cognitive delay) | follow-up phase 18 months corrected age

SECONDARY OUTCOMES:
growth in weight and head circumference | neonatal phase
time to extubation | neonatal phase
time on oxygen | neonatal phase
length of hospital stay until discharge home | neonatal phase
confirmed necrotizing enterocolitis | neonatal phase
apnea requiring treatment | neonatal phase
culture-proven infections | neonatal phase
use of post-natal steroids | neonatal phase
mean levels of hemoglobin | neonatal phase
number of transfusions | neonatal phase
number of donor exposures | neonatal phase
serum ferritin levels | neonatal phase
milder forms of cerebral palsy | follow-up phase 18 months corrected age
milder neurologic disorder | follow-up phase 18 months corrected age
personal and social functional capabilities | follow-up phase 18 months corrected age
hydrocephalus requiring a shunt | follow-up phase 18 months corrected age
seizure disorder | follow-up phase 18 months corrected age
respiratory disease | follow-up phase 18 months corrected age
iron nutritional status | follow-up phase 18 months corrected age
physical growth including head size | follow-up phase 18 months corrected age

CONTACTS AND LOCATIONS:
Overall Officials: Haresh Kirpalani, MD, MSc, Principal Investigator — McMaster University; Robin K Whyte, MD, Principal Investigator — Dalhousie University; Robin S Roberts, MTech, Study Director — McMaster University; Elizabeth Asztalos, MD, MSc, Study Director — Sunnybrook & Women's College Health Sciences Centre; Chad Andersen, MD, Study Director — Mercy Hospital for Women; Morris Blajchman, PhD, Study Director — McMaster University; Nancy Heddle, MSc, Study Director — McMaster University
Locations (10):
- United States (2):
  - Albany Medical Center, Albany, New York
  - Brooklyn Hospital Center, Brooklyn, New York
- Australia (2):
  - Royal Women's Hospital, Melbourne, Victoria
  - Mercy Hospital for Women, Melbourne, Victoria
- Canada (6):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster University, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Sunnybrook & Women's College Health Science Centre, Toronto, Ontario
  - Royal Victoria Hospital, Montreal, Quebec

REFERENCES:
- [Result] Kirpalani H, Whyte RK, Andersen C, Asztalos EV, Heddle N, Blajchman MA, Peliowski A, Rios A, LaCorte M, Connelly R, Barrington K, Roberts RS. The Premature Infants in Need of Transfusion (PINT) study: a randomized, controlled trial of a restrictive (low) versus liberal (high) transfusion threshold for extremely low birth weight infants. J Pediatr. 2006 Sep;149(3):301-307. doi: 10.1016/j.jpeds.2006.05.011. PMID 16939737
- [Result] Whyte RK, Kirpalani H, Asztalos EV, Andersen C, Blajchman M, Heddle N, LaCorte M, Robertson CM, Clarke MC, Vincer MJ, Doyle LW, Roberts RS; PINTOS Study Group. Neurodevelopmental outcome of extremely low birth weight infants randomly assigned to restrictive or liberal hemoglobin thresholds for blood transfusion. Pediatrics. 2009 Jan;123(1):207-13. doi: 10.1542/peds.2008-0338. PMID 19117884